CLINICAL TRIAL: NCT04606017
Title: Influence of Vitamin D3 Supplementation on Infliximab Efficacy in Chinese Patients With Crohn's Disease: A Retrospective Cohort Study
Brief Title: Effect of Vitamin D Supplementation on Infliximab Response in Patients With Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2020-01-213
Record Dates: First submitted 2020-10-25; First posted 2020-10-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Crohn Disease; Vitamin D Deficiency; Vitamin D Supplement
MeSH Terms: conditions — Crohn Disease; Vitamin D Deficiency | interventions — Calcium Carbonate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vitamain D: This group of patients were supplemented with 125IU/d Vitamin D
  Interventions: Drug: Caltrate Pill
- Control: The other group did not receive the supplementation of 125IU/d Vitamin D

INTERVENTIONS:
Drug: Caltrate Pill — VitD3 supplementation was defined as patients additionally took oral vitD3 (125 IU/d) within 3 days after the first infusion and persisted in the whole follow-up period.
  Groups: Vitamain D

SUMMARY:
Background: It remains uncertain whether vitD3 supplementation is beneficial for remission of Crohn's disease (CD). The influence of vitD3 supplementation on Infliximab (IFX) efficacy was retrospectively analyzed in Chinese CD patients. Methods: Patients with moderate-to-severe CD, who were bio-naïve and prescribed with IFX treatment for at least 54 weeks were recorded. VitD3 supplementation was defined as patients additionally took oral vitD3 (125 IU/d) within 3 days after the first infusion and persisted in the whole follow-up period. Disease activity was assessed using Harvey-Bradshaw Index (HBI). Serum cytokine profiles were quantitatively analyzed in a subset of all patients at baseline and 54-week after intervention.

ELIGIBILITY:
Inclusion Criteria:

* moderate-to-severe CD
* Treated with Infliximab
* bio-naïve at the time of diagnosis

Exclusion Criteria:

* had recent supplementation of vitD3
* had prior or concomitant use of other biologic agent, glucocorticoid and/or immunomodulators at the time of enrollment
* pregnant
* had cognitive/developmental disorders that affected their ability to complete the study procedures
* had medical illness or therapies potentially affecting bone, nutrition or growth status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Serum 25 (OH) D level | 54 weeks
  Because serum 25 (OH) D levels are relatively stable, they are considered the most reliable indicator of vitamin D status.
disease activity | 54 weeks
  CDAI evaluation

SECONDARY OUTCOMES:
the metabolism of calcium and phosphorus | 54 weeks
  serum levels calcium and phosphorus
the expression profiles of Th-cell-related cytokines | 54 weeks
  Serum levels of IL-2, IL-4, IL-6, IL-10, TNF-α and IFN-γ

CONTACTS AND LOCATIONS:
Overall Officials: Xia sheng long long, Master, Study Director — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- SAHWenzhouMU, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
Data sets will be made available on relevant requests and in accordance with journal guidelines when publishing results from this study.

REFERENCES:
- [Derived] Xia SL, Min QJ, Shao XX, Lin DP, Ma GL, Wu H, Cao SG, Jiang Y. Influence of Vitamin D3 Supplementation on Infliximab Effectiveness in Chinese Patients With Crohn's Disease: A Retrospective Cohort Study. Front Nutr. 2021 Oct 22;8:739285. doi: 10.3389/fnut.2021.739285. eCollection 2021. PMID 34746207